CLINICAL TRIAL: NCT04577625
Title: A Double-blind Randomized Clinical Study Investigating Lactobacillus Reuteri Supplementations Influence on Testosterone Levels in Healthy Men
Brief Title: Effect of Probiotics on Testosterone in Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioGaia AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CSUB0176
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2020-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- L. reuteri Low Dose (Active Comparator): L. reuteri will be delivered in a capsule at a low dose including Vitamin D3. Administration twice daily.
  Interventions: Dietary Supplement: Lactobacillus reuteri (L. reuteri)
- L. reuteri High Dose (Active Comparator): L. reuteri will be delivered in a capsule at a high dose including Vitamin D3. Administration twice daily.
  Interventions: Dietary Supplement: Lactobacillus reuteri (L. reuteri)
- Placebo (Placebo Comparator): The placebo product will be identical to the active product in taste and appearance and include Vitamin D3 but without the L. reuteri. Administration twice daily.
  Interventions: Dietary Supplement: Lactobacillus reuteri (L. reuteri)

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri (L. reuteri) — L.reuteri high or low dose with vitamin D3 compared to vitamin D3 only

SUMMARY:
This study evaluates the effect of L. reuteri ATCC PTA 6475 supplementation on testosterone in men.

DETAILED DESCRIPTION:
The probiotic Lactobacillus reuteri ATCC PTA 6475 has been shown to modulate testosterone levels in mice. It is not known if these effects are seen in humans and this trial is intended to study this.

The aim of this study is to investigate if L. reuteri ATCC PTA 6475 will effect blood testosterone levels in in healthy male subjects 50-65 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give signed informed consent for participation in the study.
* Healthy males aged between 50-65 with no known underlying medical conditions
* Subjects who are capable of taking themselves to testing centre at 3 separate timepoints (Baseline, week 6 and week 12).
* Subjects who are available to give fasting blood samples before 10am on day of blood sample collection
* No history of androgen or testosterone supplementation within 6 months prior to study start.
* Subjects who have not been taking antibiotics or probiotic supplements 4 weeks prior to study start 8. Able and willing to comply with the restirictions defined for the study period
* Ability to understand and comply with the requirements of the study, as judged by the investigator physician

Exclusion Criteria:

* Subjects who presently have or have had cardiovascular issues in the past 2 years.
* Subjects who have a Body Mass Index of < 18 or > 30
* Known elevated Prostate Specific Antigen levels.
* History of prostate or testicular cancer.
* Nicotine abuse
* Alcohol abuse

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2021-06-05 (Actual)

PRIMARY OUTCOMES:
Concentration of total testosterone | Baseline, 6 weeks, 12 weeks
  Change in total testosterone concentration over time

SECONDARY OUTCOMES:
Free testosterone index | Baseline, 6 weeks, 12 weeks
  Change in Free testosterone index (100x(Testosterone/SHBG) over time
Percentage of hematokrit | Baseline, 6 weeks, 12 weeks
  Change in Hematokrit over time
Number of adverse events | Continously 12 weeks
  Adverse event from administration of first dose until 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Health & Society, Malmö University, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided